CLINICAL TRIAL: NCT03597295
Title: A Phase 2 Study of INCMGA00012 in Participants With Squamous Carcinoma of the Anal Canal Who Have Progressed Following Platinum-Based Chemotherapy (POD1UM-202)
Brief Title: A Study of INCMGA00012 in Squamous Carcinoma of the Anal Canal Following Platinum-Based Chemotherapy (POD1UM-202)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCMGA 0012-202; 2018-002070-51 (EudraCT Number)
Record Dates: First submitted 2018-07-16; First posted 2018-07-24 (Actual); Results first posted 2021-08-23 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Squamous Cell Carcinoma of Anal Canal
Keywords: Squamous carcinoma of the anal canal; anti-PD-1 antibody; IgG4 monoclonal antibody; INCMGA00012

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Retifanlimab 500 mg (Experimental): Retifanlimab 500 milligrams (mg) intravenously every 4 weeks (Q4W).
  Interventions: Drug: Retifanlimab

INTERVENTIONS:
Drug: Retifanlimab — Retifanlimab 500 milligrams (mg) intravenously every 4 weeks (Q4W).
  Other Names: MGA012; INCMGA00012

SUMMARY:
The purpose of this study is to assess the efficacy of INCMGA00012 in participants with locally advanced or metastatic squamous carcinoma of the anal canal (SCAC) who have progressed after platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written informed consent form.
* Confirmed diagnosis of locally advanced or metastatic SCAC.
* Must have received (or been intolerant to or ineligible for) at least 1 prior line of platinum-based chemotherapy and received no more than 2 prior systemic treatments.
* Must have measurable disease by RECIST v1.1.
* Eastern Cooperative Oncology Group performance status of 0 to 1.
* If HIV-positive, then all of the following criteria must also be met: CD4+ count ≥ 300/μL, undetectable viral load, and receiving highly active antiretroviral therapy.

Exclusion Criteria:

* Receipt of anticancer therapy or participation in another interventional clinical study within 21 days before the first administration of study drug; 6 weeks for mitomycin C.
* Radiotherapy within 14 days of first dose of study treatment with the following caveats: 28 days for pelvic radiotherapy, 6 months for thoracic region radiotherapy that is > 30 Gy.
* Prior treatment with programmed cell death protein 1 (PD-1) or programmed cell death ligand protein 1 (PD-L1)-directed therapy.
* Active autoimmune disease requiring systemic immunosuppression.
* Known central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Known active hepatitis infection.
* Active infections requiring systemic therapy.
* Is pregnant or breastfeeding or is expecting to conceive or father children within the projected duration of the study, from screening through 6 months after the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2021-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (46):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - Maryland Oncology Hematology P.A., Rockville, Maryland
  - Texas Oncology-Baylor Charles A. Sammons, Dallas, Texas
  - Texas Oncology-McKinney, McKinney, Texas
  - Renovatio Clinical, Spring, Texas
- Belgium (2):
  - Zna Middelheim, Antwerp
  - Hopital Erasme, Brussels
- Denmark (3):
  - Aarhus Universitets Hospital, Aarhus
  - Herlev Og Gentofte Hospital, Herlev
  - Vejle Hospital, Vejle
- France (7):
  - Centre Hospitalier Universitaire de Besancon, Besançon
  - CHU Hopital De La Timone, Marseille
  - Icm Montpellier, Montpellier
  - Hopital Universitaire Pitie-Salpetriere, Paris
  - Chu de Rennes - Hôpital Pontchaillou, Rennes
  - Centre de Lutte Contre Le Cancer - Institut de Cancerologie de L'Ouest - Rene Gauducheau, Saint-Herblain
  - CHU Toulouse Hopital Rangueil, Toulouse
- Germany (2):
  - University Medical Centre Hamburg-Eppendorf, Centre of Oncology, Hamburg
  - Asklepios Klinik Altona, Hamburg
- Italy (10):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Ancona
  - Ospedale A. Perrino - Brindisi, Brindisi
  - A.O.U. Policlinico V. Emanuele G. Rodolico, Catania
  - Ospedale Degli Infermi - Faenza, Faenza
  - Irccs Azienda Ospedaliera Universitaria San Martino, Genova
  - Niguarda Cancer Center, Milan
  - Aou Modena - Policlinico, Modena
  - Clinica La Maddalena, Palermo
  - Policlinico Universitario Agostino Gemelli Universita Cattolica Del Sacro Cuore, Rome
  - IRCCS Casa Sollievo Della Sofferenza, San Giovanni Rotondo
- Norway (2):
  - Haukeland U Hospital Bergen, Bergen
  - Oslo U, Oslo
- Spain (3):
  - Hospital General Universitari Vall D Hebron, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (10):
  - Royal Sussex County Hospital, Brighton
  - Royal Marsden Hospital, Chelsea
  - Castle Hill Hospital, Cottingham
  - St. James U Hospital, Leeds
  - St. James Univ Hospital, Leeds
  - Royal Free London Nhs Foundation Trust, London
  - The Royal Marsden Nhs Foundation Trust - Chelsea, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Marsden Hospital, Sutton
  - Royal Cornwall Hospital, Sunrise Centre, Truro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rao S, Anandappa G, Capdevila J, Dahan L, Evesque L, Kim S, Saunders MP, Gilbert DC, Jensen LH, Samalin E, Spindler KL, Tamberi S, Demols A, Guren MG, Arnold D, Fakih M, Kayyal T, Cornfeld M, Tian C, Catlett M, Smith M, Spano JP. A phase II study of retifanlimab (INCMGA00012) in patients with squamous carcinoma of the anal canal who have progressed following platinum-based chemotherapy (POD1UM-202). ESMO Open. 2022 Aug;7(4):100529. doi: 10.1016/j.esmoop.2022.100529. Epub 2022 Jul 8. PMID 35816951

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 40 study centers: 32 in France, 19 in the United Kingdom, 10 in Italy, 10 in Spain, 7 in Denmark, 6 in the United States, 4 in Norway, 4 in Belgium, and 2 in Germany.
Pre-assignment Details: A total of 94 participants with locally advanced or metastatic squamous carcinoma of the anal canal were enrolled in the study and treated with retifanlimab.
Groups:
- Retifanlimab 500 mg: Participants received retifanlimab 500 milligrams (mg) intravenously every 4 weeks (Q4W).
Period: Overall Study
Arm/Group | Retifanlimab 500 mg
Started | 94
Completed | 17
Not Completed | 77
Not completed — Death | 70
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants enrolled in the study who received at least 1 dose of study drug.
Units Other Than Participants: 94
Arm/Group | Retifanlimab 500 mg
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.1 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 49
  Not Reported | 33
  Unknown | 4
  Missing | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 72
  Black/African-American | 1
  Captured as "Other" | 4
  Missing | 6
  Not Reported | 11

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR), per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1), as assessed by independent central radiographic (ICR) review, at any post-Baseline visit until new anti-cancer therapy or first Progressive Disease. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: Cycle 1 Day 1, and every 4 weeks throughout the study, up to approximately 24 months
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Retifanlimab 500 mg
Number analyzed (Participants) | 94
percentage of participants | 13.8

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from an initial objective response (CR or PR) per RECIST v1.1 until the first observation of documented disease progression (PD), as determined by ICR, or death due to any cause. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion.
Time Frame: up to 18.2 months
Population: Full Analysis Set. All participants with confirmed tumor responses (CR or PR) by ICR according to RECIST v1.1 were analyzed. The 95% confidence interval was calculated using the Brookmeyer and Crowley's method and Klein and Moeschberger's method with log-log transformation.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Retifanlimab 500 mg
Number analyzed (Participants) | 13
months | 9.5 [4.4 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with a confirmed overall response of CR, PR, or stable disease (SD), per RECIST v1.1, at any post-baseline visit until the first progressive disease (PD) or new anti-cancer therapy. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion. SD: no change in target lesions to qualify for CR, PR, or PD.
Time Frame: Cycle 1 Day 1, and every 4 weeks throughout the study, up to approximately 24 months
Population: Full Analysis Set. Confidence intervals were calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Retifanlimab 500 mg
Number analyzed (Participants) | 94
percentage of participants | 48.9 [38.5 to 59.5]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: According to RECIST 1.1, PFS was defined as the length of time from the initial infusion of study drug until the earliest date of disease progression, as determined by ICR, or death due to any cause, if occurring sooner than progression.
Time Frame: up to 16.8 months
Population: Full Analysis Set. Median PFS time was estimated using the Kaplan-Meier method. The confidence interval for median PFS time was calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Retifanlimab 500 mg
Number analyzed (Participants) | 94
months | 2.3 [1.9 to 3.6]

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time in months between the first dose date (Day 1) and the date of death due to any cause.
Time Frame: up to 28.2 months
Population: Full Analysis Set. Median survival time was estimated using the Kaplan-Meier method. The confidence interval for median survival time was calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Retifanlimab 500 mg
Number analyzed (Participants) | 94
months | 13.4 [10.1 to 15.0]

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of the study drug. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of retifanlimab and within 90 days of the last administration of retifanlimab.
Time Frame: up to 913 days
Population: Safety Evaluable Population: all enrolled participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Retifanlimab 500 mg
Number analyzed (Participants) | 94
Participants | 90

7. Secondary Outcome: Cmax of Retifanlimab
Description: Cmax was defined as the maximum observed plasma concentration.
Time Frame: pre-infusion on Day 1 of Cycles 1, 2, 4, 6, and 7; 10 minutes and 4 hours post-infusion on Day 1 of Cycles 1 and 6
Population: Pharmacokinetic (PK) Evaluable Population: all participants who received at least 1 dose of study drug and provided a Baseline and at least 1 postdose serum sample (1 PK measurement)
Measure: Mean (Standard Deviation); unit: milligrams per Liter (mg/L)
Arm/Group | Retifanlimab 500 mg
Number analyzed (Participants) | 92
milligrams per Liter (mg/L) | 151 (27.6)

8. Secondary Outcome: Tmax of Retifanlimab
Description: tmax was defined as the time to the maximum concentration.
Time Frame: pre-infusion on Day 1 of Cycles 1, 2, 4, 6, and 7; 10 minutes and 4 hours post-infusion on Day 1 of Cycles 1 and 6
Population: PK Evaluable Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Retifanlimab 500 mg
Number analyzed (Participants) | 92
hours | 1.20 (0.305)

9. Secondary Outcome: Cmin of Retifanlimab
Description: Cmin was defined as the minimum observed plasma concentration over the dose interval.
Time Frame: pre-infusion on Day 1 of Cycles 1, 2, 4, 6, and 7; 10 minutes and 4 hours post-infusion on Day 1 of Cycles 1 and 6
Population: PK Evaluable Population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Retifanlimab 500 mg
Number analyzed (Participants) | 92
mg/L | 22.4 (7.87)

10. Secondary Outcome: AUC0-t of Retifanlimab
Description: AUC0-t was defined as the area under the plasma concentration-time curve from time = 0 to the last measurable concentration at time = t.
Time Frame: pre-infusion on Day 1 of Cycles 1, 2, 4, 6, and 7; 10 minutes and 4 hours post-infusion on Day 1 of Cycles 1 and 6
Population: PK Evaluable Population
Measure: Mean (Standard Deviation); unit: day*mg/L
Arm/Group | Retifanlimab 500 mg
Number analyzed (Participants) | 92
day*mg/L | 1950 (594)

ADVERSE EVENTS:
Time Frame: up to 913 days
Description: Treatment-emergent adverse events (TEAEs), defined as any AEs either reported for the first time or the worsening of pre-existing events after the first dose of retifanlimab and within 90 days of the last administration of retifanlimab, have been reported.
Arm/Group | Retifanlimab 500 mg
All-Cause Mortality (participants affected / at risk) | 60/94
Serious Adverse Events (participants affected / at risk) | 50/94
Other Adverse Events (participants affected / at risk) | 79/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retifanlimab 500 mg (N=94)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Anal abscess (Infections and infestations) | 1 (1)
Asthenia (General disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Body temperature increased (Investigations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Catheter site pain (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 1 (1)
Coma hepatic (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
General physical health deterioration (General disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1)
Inadequate analgesia (General disorders) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Lyme disease (Infections and infestations) | 1 (1)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (4)
Pain (General disorders) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pelvic infection (Infections and infestations) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 3 (3)
Peritonitis (Infections and infestations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 2 (3)
Proctitis haemorrhagic (Gastrointestinal disorders) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Stoma site infection (Infections and infestations) | 1 (1)
Superior mesenteric artery syndrome (Gastrointestinal disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ureteric compression (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4)
Venous thrombosis limb (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retifanlimab 500 mg (N=94)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Anaemia (Blood and lymphatic system disorders) | 15 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (10)
Aspartate aminotransferase increased (Investigations) | 7 (7)
Asthenia (General disorders) | 22 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9)
Constipation (Gastrointestinal disorders) | 12 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (13)
Cystitis (Infections and infestations) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 12 (12)
Diarrhoea (Gastrointestinal disorders) | 20 (32)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (13)
Fatigue (General disorders) | 17 (21)
Headache (Nervous system disorders) | 8 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5)
Hypothyroidism (Endocrine disorders) | 9 (10)
Insomnia (Psychiatric disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 15 (21)
Proctalgia (Gastrointestinal disorders) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (14)
Pyrexia (General disorders) | 10 (18)
Rash (Skin and subcutaneous tissue disorders) | 5 (6)
Rectal haemorrhage (Gastrointestinal disorders) | 9 (17)
Urinary tract infection (Infections and infestations) | 7 (9)
Vomiting (Gastrointestinal disorders) | 14 (18)
Weight decreased (Investigations) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT03597295/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT03597295/SAP_001.pdf